CLINICAL TRIAL: NCT06866314
Title: Comparison of VitalPLANT and Helichrysum Italicum Infusions Effects on the Components of Metabolic Syndrome in Adults
Brief Title: Clinical Trials of VitalPLANT and Helichrysum Infusions in Adults ( VitalPlant_SMILJ )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Institute of food technology Novi Sad (Unknown); Josip Pančič Institute Belgrade (Unknown)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate Professor, PhD, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: VitalPLANT and SMILJ_clinical
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Metabolic Syndrome
Keywords: functional food; tea infusion; overweight; metabolic syndrome
MeSH Terms: conditions — Overweight; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VitalPLANT (Active Comparator): 0.75 g of milled plant material (VitalPLANT)
  Interventions: Dietary Supplement: Tea infusion VitalPLANT - Active comparator
- VitalPLANT+Helichrysum Italicum (Experimental): 0.75 g of milled plant material (VitalPLANT) + 0.75 g of milled Helichrysum Italicum
  Interventions: Dietary Supplement: Tea infusion VitalPLANT + Helichrysum Italicum - Experimental product

INTERVENTIONS:
Dietary Supplement: Tea infusion VitalPLANT - Active comparator — Consumation of 200 mL of tea infusion (VitalPLANT) in the morning 30 min before breakfast for one week
  Arms: VitalPLANT
Dietary Supplement: Tea infusion VitalPLANT + Helichrysum Italicum - Experimental product — Consumation of 200 mL of tea infusion VitalPLANT + Helichrysum Italicum in the morning 30 min before breakfast for one week
  Arms: VitalPLANT+Helichrysum Italicum

SUMMARY:
The study evaluates the effects of VitalPLANT and Helichrysum italicum on different components of the metabolic syndrome. The components of metabolic syndrome will be measured at baseline and one week after daily consumption of either VitalPLANT alone or either VitalPLANT+Helichrysum italicum after one week of washout.

DETAILED DESCRIPTION:
"VITALPLANT" medicinal plant mixture, aimed at body weight regulation and metabolism enhancement was formulated in order to be incorporated as an ingredient in functional food formulations on the basis of known biological activity of the alder buckthorn bark, peppermint, caraway and parsley. Medicinal plants have long been known as sources of biologically active substances.Oil component apiole - a proven kidney stimulant and parsley (Petroselinum crispum (Mill.) A.W. Nym. ex Hill) are known for their diuretic action. Peppermint (Mentha x piperita L.) and caraway (Carum Carvi L.) essential oils are frequently used in herbal drugs for treatment of abdominal discomfort and pain, while the alder buckthorn bark (Rhamnus Frangula L.) contains anthraquinone glycosides with purgative effects. "Vitalplant" mixture was found to be beneficial for the reduction of body weight and improvement of antioxidant status of the erythrocytes, and its antihyperlipidemic property was highly active for enhancing the profile of plasma lipids in rats.

Similarly, Helichrysum italicum (HI) is also widely used in traditional medicine. Lately, it has been shown that HI infusion consumption had a beneficial effect on anthropometric traits. Indeed, significant reductions in body weight, body mass index, and visceral and total body fat were observed in adults. Moreover, after four weeks of intervention, LDL decreased and serum antioxidant properties were improved. Therefore, consuming infusion could thus be recommended as a simple, profitable habit for individuals with traits of metabolic syndrome.

Therefore, the aim of our study is to evaluate the effects of VitalPLANT alone and VitalPlant+Helichrysum italicum on different components of the metabolic syndrome in adults presenting at least two components of metabolic syndrome and yet not receiving any medication. The components of metabolic syndrome (lipid profile, blood pressure, antrophometry, inflammation status, glucose levels) will be measured at baseline and one week after daily consumptions of either VitalPLANT alone or VitalPLANT+SMILJ. In between there will be one week of washout period.

ELIGIBILITY:
Inclusion Criteria:

* stable weight in the last 3 months
* BMI more than 25
* clinical diagnosis of at least two components of metabolic syndrome

Exclusion Criteria:

* consumption of dietary supplements
* medications for any component of metabolic syndrome

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Body weight | changes from baseline to one week of daily consumption of VitalPLANT alone, after one week washout and after one week of daily consumption of VitalPLANT+SMILJand after two weeks of washout
  Changes in body weight (in kilograms) will be examined with bioelectrical impedance analysis (BIA) Tanita MC-980MA (Maeno-cho, Japan) and dedicated software (GMON Pro-Tanita)

SECONDARY OUTCOMES:
Anthropometric measurements | changes from baseline to one week of daily consumption of VitalPLANT alone, after one week washout and after one week of daily consumption of VitalPLANT+SMILJand after two weeks of washout
  Changes in body fat (in kilograms and %) will be examined with bioelectrical impedance analysis (BIA) Tanita MC-980MA (Maeno-cho, Japan) and dedicated software (GMON Pro-Tanita).
Lipid profile | changes from baseline to one week of daily consumption of VitalPLANT alone, after one week washout and after one week of daily consumption of VitalPLANT+SMILJand after two weeks of washout
  Changes in total cholesterol, LDL cholesterol, HDL cholesterol and triacylglycerides will be examined with biochemical analyzer Cobass
nflammation | changes from baseline to one week of daily consumption of VitalPLANT alone, after one week washout and after one week of daily consumption of VitalPLANT+SMILJand after two weeks of washout
  Changes in C-reactive protein levels will be examined with biochemical analyzer Cobass
Glucose levels | changes from baseline to one week of daily consumption of VitalPLANT alone, after one week washout and after one week of daily consumption of VitalPLANT+SMILJand after two weeks of washout
  Changes in glucose levels will be examined with biochemical analyzer Cobass

CONTACTS AND LOCATIONS:
Overall Officials: Zala Jenko Pražniakr, phD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University Of Primorska Faculty of Health Sciences, Izola, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No